CLINICAL TRIAL: NCT00003727
Title: Autotransplantation for Chronic Myelogenous Leukemia (CML) Followed by Immunotherapy With Ex-Vivo Expanded Autologous T Cells
Brief Title: Chemotherapy and Peripheral Stem Cell Transplantation Followed by Immunotherapy in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066839; MSGCC-9851; MSGCC-1198006; NCI-V98-1513
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia; Philadelphia chromosome negative chronic myelogenous leukemia; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Filgrastim; Interferon-alpha; sargramostim; Carmustine; Cyclophosphamide; Etoposide; Gemcitabine; Melphalan

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Biological: sargramostim
Biological: therapeutic autologous lymphocytes
Drug: carmustine
Drug: cyclophosphamide
Drug: etoposide
Drug: gemcitabine hydrochloride
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with a peripheral stem cell transplant and immunotherapy may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: This phase II trial is studying giving chemotherapy together with a peripheral stem cell transplant followed by immunotherapy to see how well it works in treating patients with chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of ex vivo expansion and reinfusion of autologous CD4+ T cells after interferon therapy or high-dose chemotherapy with CD34-selected autologous peripheral blood stem cell rescue in patients with chronic phase chronic myelogenous leukemia (CML).
* Determine the frequency of hematologic, cytogenetic, and molecular remissions of CML following infusion of ex vivo expanded T cells.

OUTLINE: Patients undergo mononuclear cell leukapheresis to obtain T cells for ex-vivo expansion, preferably before they receive interferon alfa subcutaneously (SC) daily on a therapeutic trial.

At least 1 month after interferon is stopped, mobilization chemotherapy is administered. Patients receive cyclophosphamide IV over 12 hours on day 0, etoposide IV over 2 hours on day 1, sargramostim (GM-CSF) SC on days 3 and 4, and filgrastim (G-CSF) SC beginning on day 5. Peripheral blood stem cells (PBSC) are collected by leukapheresis when blood cell counts have recovered.

Approximately 2-3 weeks later, high-dose chemotherapy begins. Patients receive gemcitabine IV over 100 minutes on day -5, carmustine IV over 2 hours on day -2, followed 6 hours later by gemcitabine IV again, and melphalan IV over 20 minutes on day -1. CD34 selected PBSCs are infused on day 0, at least 18 hours after melphalan administration. Patients receive GM-CSF SC beginning on day 1 and continuing until blood cell counts recover.

Patients then receive ex vivo expanded autologous T cells on day 14 after autotransplantation. Interferon alfa is administered three times a week starting about 3 months after transplantation.

Patients who only receive expanded T cells, without high-dose chemotherapy and autotransplantation, but show no response after 3 months, may proceed to autotransplantation followed by a second ex vivo expanded T-cell infusion.

Patients are followed at 1, 2, 3, 6, 9, and 12 months, then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 7-22 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myelogenous leukemia based on clinical features and molecular evidence for bcr/abl gene rearrangement

  * First or second chronic phase at the time of stem cell collection
* Ineligible for allogeneic transplantation
* Should receive interferon alfa (IFN-A) with or without low-dose cytarabine for at least 3-6 months before autotransplantation and meet one of the following conditions:

  * After 3 months of IFN-A, hematologic response is partial or less and poor clinical feature was present at diagnosis
  * After 6 months of IFN-A, hematologic response is partial or complete (but 100% Ph+) and poor clinical feature was present at diagnosis
  * After 9 or 12 months of IFN-A, no cytogenetic response occurred (100% Ph+), regardless of pretreatment clinical features
  * After at least 12 months of IFN-A (or on 2 separate tests, 3 months apart), only minor cytogenetic response (35-90% Ph+) occurred, then eligible for ex vivo expanded autologous T cells only (without high-dose chemotherapy or autografting) or high-dose therapy plus autographing at physicians' discretion
  * After at least 12 months of IFN-A (or on 2 tests, 3 months apart), major but not complete cytogenetic response (0-34% Ph+) occurred, then eligible for ex vivo expanded autologous T cells only (without high-dose chemotherapy or autografting)
  * After at least 18 months of IFN-A, complete cytogenetic response (0% Ph+) occurred but remain positive for BCR/ABL gene rearrangement then eligible for ex vivo expanded autologous T cells only (without high-dose chemotherapy or autografting)
* Unsatisfactory response to prior STI571 allowed (regardless of prior IFN-A)

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN) (unless due to Gilbert's disease)
* AST and ALT no greater than 2 times ULN (unless liver involvement with CML)

Renal:

* Creatinine no greater than 2.5 mg/dL

Cardiovascular:

* LVEF at least 45% (lower allowed if no significant functional impairment)

Pulmonary:

* FEV_1, FVC, and DLCO at least 50% predicted

Other:

* No active infections requiring IV antibiotics
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 1 month since prior interferon

Chemotherapy:

* At least 1 week since hydroxyurea before leukapheresis

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 1999-03; Primary Completion 2005-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Response (i.e., major cytogenetic or molecular response) within 12 months after completion of study therapy
Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P. Rapoport, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland, United States